CLINICAL TRIAL: NCT04301960
Title: Comparison of the Effects of Single and Dual Task Training on Processing Speed, Cognitive Functions, Walking Speed, Dual Task Performance and Balance Functions in Individuals With Mild Cognitive Impairment
Brief Title: Effects of Single and Dual Task Training in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Betül Fatma Bilgin, Research assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/23-11
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Single-task; Dual-task; Processing Speed; Cognitive Functions; Walking Speed; Balance Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single task group (Experimental): The single task group includes balance gaining and cognitive training. The single task group will have 30-40 minutes of single-task training for 3 sessions per week for 8 weeks.
  Interventions: Other: Single task training
- Dual-task (Experimental): The dual-task group includes CSRT Mat training. The dual-task group will have CSRT Mat training for 30-40 minutes of dual-task training for 3 sessions per week for 8 weeks.
  Interventions: Other: Dual task training

INTERVENTIONS:
Other: Single task training — The single task group includes balance gaining and cognitive training. The single task group will have 30-40 minutes of single-task training for 3 sessions per week for 8 weeks.
  Arms: Single task group
Other: Dual task training — The dual-task group includes CSRT Mat training. The dual-task group will have CSRT Mat training for 30-40 minutes of dual-task training for 3 sessions per week for 8 weeks.
  Arms: Dual-task

SUMMARY:
The aim of this study is to compare the effects of single and dual-task training on processing speed, cognitive functions, walking speed, dual-task performance and balance functions in individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is a cognitive impairment that usually occurs with the normal cognitive decline with age and does not significantly affect daily function. MCI is diagnosed by the presence of one or more cognitive deficits that occur without meeting the diagnostic criteria of dementia. MCI is regarded as an intermediate stage between normal cognition and dementia. Also known as the early stage of dementia. Although 6 main cognitive domains could potentially be affected (learning and memory, social functioning, language, visuospatial function, complex attention, or executive functioning), the term "mild cognitive impairment" generally refers to a decline in the ability to learn new information or recall stored information. While the current dementia criteria require that cognitive functions be impaired to prevent an individual from continuing his/her daily life independently, MCI is the stage where there is no significant problem in the daily life of the individual before this stage. Risk factors include male sex, presence of the apolipoprotein E allele, family history of cognitive impairment, and the presence of vascular risk factors such as hypertension, hyperlipidemia, coronary artery disease, and stroke.

Training of cognitive functions with physiotherapy can be effective in improving various aspects of objective cognitive functioning (memory performance, executive functioning, processing speed, attention, fluid intelligence, and subjective cognitive performance). It has been reported that there is a slowdown or decrease in cognitive status through training. In the literature, there were no studies comparing single and dual-task training effects in patients with mild cognitive impairment. Therefore, the aim of this study is to compare the effects of single and dual-task training on the processing speed, cognitive functions, walking speed, dual-task performance and balance functions in individuals with mild cognitive impairment.

Participants who are between the ages of 65-85, who has Montreal Cognitive Assessment score between 13-26, the Quick Mild Cognitive Impairment Screen score between 48-67, Instrumental Activities of Daily Living Scale score ≥6/8, who says yes to "Do you have a memory problem?", who can walk independently without using any walking aids and who are likely to be MCI as a result of the tests will be referred to the neurologist and those whose diagnosis is confirmed will be included in this study. Participants who have any musculoskeletal disorders that may cause balance and gait disorders, central or peripheral neurological diseases (eg. stroke, Parkinson's disease or polyneuropathies), using psychiatric drugs that may affect psychiatric disease and / or cognitive performance, daltonism diagnosed and who attending any exercise program will not be included in this study.

All the participants will be measured with Choice Stepping Reaction Time (CSRT) Test, Stroop Test, backward counting, verbal fluency, 10 meters walking test (10MWT), 10MWT with backward counting and verbal fluency for dual tasking, Fullerton Advanced Balance (FAB) Scale and D+R Balance Application. The measurements will be made at the beginning of the treatment (0 week) and at the end of the treatment (8 weeks).

The choice stepping reaction time (CSRT) task has been better to discriminate between fallers and non-fallers than other sensorimotor and balance measures and to predict falls in older people, mediated through physiologic and cognitive pathways.

The single task group includes balance gaining and cognitive training. In the dual-task group includes CSRT Mat training.

The single task group will have 30-40 minutes of single-task training for 3 sessions per week for 8 weeks. The dual-task group will have CSRT Mat training for 30-40 minutes of dual-task training for 3 sessions per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are between 65-85 years of age,
2. Who has the Montreal Cognitive Assessment score between 13-26,
3. Who has the Quick Mild Cognitive Impairment screen score between 48-67,
4. Who has Instrumental Activities of Daily Living Scale score ≥6/8,
5. Who says yes to "Do you have a memory problem?" question,
6. Who can walk independently without using any walking aids and
7. Who is likely to have mild cognitive impairment as a result of the tests will be referred to the neurologist and those whose diagnosis is confirmed will be included in this study.

Exclusion Criteria:

1. Participants who have any musculoskeletal disorders that may cause balance and gait disorders,
2. Who have central or peripheral neurological diseases (eg. stroke, Parkinson's disease or polyneuropathies),
3. Who are using psychiatric drugs that may affect psychiatric disease and/or cognitive performance,
4. Who has daltonism and
5. Who attends any exercise program will not be included in this study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Choice Stepping Reaction Time Test (CSRT) | 8 weeks
  A custom-made Choice Stepping Reaction Time step pad (CSRT-MAT) and a computer unit will be used to evaluate the processing speed. The system is consisted of a CSRT-MAT having pressure-sensitive panels and a display monitor connected to a computer unit. The computer unit recorded the timing of foot lift and landing. The step direction is indicated by one arrow changing its color. The CSRT device included 2 tests: Stepping Reaction Time (SRT) and Stroop Test (ST). In this study, only the SRT test will be done. In the SRT test, the participants are asked to step as quickly as possible onto the corresponding arrow on the CSRT-MAT and then return to the center. The reaction time (RT) measured from stimulus occurrence to movement initiation (lift off), movement time (MT) measured from movement initiation to step finalization (step down) and total response time (RsT) measured as the sum of RT and MT.

SECONDARY OUTCOMES:
Stroop Test | 8 weeks
  The Stroop Color and Word Test (SCWT) will be used to assess selective attention. SCWT is a neuropsychological test extensively used for both experimental and clinical purposes. It assesses the ability to inhibit cognitive interference, which occurs when the processing of a stimulus feature aﬀects the simultaneous processing of another attribute of the same stimulus. Named color-word (CW) condition, color-words are printed in an inconsistent color ink (for instance the word "red" is printed in green ink). Thus, in this incongruent condition, participants are required to name the color of the ink instead of reading the word. At the completion of the test, the number of incorrect responses and time of completion scores will be recorded. The test has a total of 50 questions and the application takes approximately 5 minutes.
Verbal Fluency Test (VFT) | 8 weeks
  The Verbal Fluency Test (VFT) will be used to evaluate the verbal fluency ability of the participants. Verbal fluency is the ability to generate an appropriate strategy for word searching. The test consists of giving the person 1 minute to verbally list as many things as possible in a category. The verbal fluency test will be done in two different ways. The first one is semantic subtest, in this test the words are generated according to a category (such as 'animals' or 'fruits'). The other one is the phonological fluency subtest, in this test participants are asked to generate words according to the letter they begin with (such as 'F', 'A' or 'S') and on semantic fluency. The correct number of answers within 1 minute will be determined after the completion of the test by listening to voice recorder recordings.
Serial Subtraction Test (SST) | 8 weeks
  The Serial Subtraction Test (SST) will be used to evaluate the arithmetic performance and mental tracking capacity of the participants. Counting backward is thought to be a simple mental tracking task, which requires the subject to hold information regarding a tracking number in mind while subsequently reversing the order of a set of numbers. The failure to count backward is likely caused by an intrusion of the inappropriate routine schema (e.g. the process of counting forward), as the process of counting forward is more acquired and automatic than that of counting backward. Therefore the investigators preferred to use the counting backward in this study. In this test, the participants will be asked to "subtract 7 from 100" (Serial 7s) and to keep going until they can't go any further".
10 Meter Walking Test (10 MWT) | 8 weeks
  The 10 Meter Walk Test (10 MWT) is a performance measure used to assess walking speed in meters per second over a short distance. In 10 MWT individuals walk (at a normal pace) without assistance for 10 meters and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration. The timing is started when the toes of the leading foot cross the 2-meter mark and stoped at the 8-meter mark. The total time taken to ambulate 6 meters will be recorded and then divided by the total time (in seconds) in m/s.
10 Meter Walking Test with Verbal Fluency Test (10 MWT-VFT) | 8 weeks
  The 10 Meter Walking Test with verbal fluency test (10 MWT-VFT) will be used to evaluate the dual-task (motor and cognitive) skills of the participants. In the 10 MWT-VFT, the participants will be evaluated during both conditions: verbal fluency and 10 MWT. While the patients are walking in they will be counting verbally as many things as possible in a category. The correct number of answers while walking will be determined after the completion of the test by listening to voice recorder recordings.
10 Meter Walking Test with Serial Subtraction Test (10 MWT-SST) | 8 weeks
  The 10 Meter Walking Test with Serial Subtraction Test (10 MWT-SST) will be used to evaluate the dual-task (motor and cognitive) skills of the participants. In the 10 MWT-SST the participants will be evaluated during both conditions: serial subtraction and 10 MWT. While the patients are walking in they will be asked to "subtract 7 from 100" (Serial 7s) and to keep going until they can't go any further". The correct number of answers while walking will be determined after the completion of the test by listening to voice recorder recordings.
Fullerton Advanced Balance (FAB) Scale | 8 weeks
  The Fullerton Advanced Balance (FAB) scale will be used to evaluate the balance performance of the participants. This performance-based scale consists of 10 test items assessing functional balance (static and dynamic) status. The individual test items are feet together, eyes closed (1), reach forward to retrieve an object (2), turn in a full circle (3), step up and over a bench (4), tandem walk (5), stand on one leg (6), stand on foam, eyes closed (7), two-footed jump (8), walk with head turns (9) and reactive postural control (10). Each test item is scored using a 0-4 scale. The highest score is 40 points, and the lowest is zero. Higher scores indicate better balance abilities. The FAB scale is quick to administer (∼10-12 min) and can be administered in a relatively small area.
D+R Balance Application | 8 weeks
  The D+R Balance Application of iPhone will be used to evaluate the postural sway of the participants. The iPhone will be inserted into an incase armband and will be strapped to the participant's right upper arm. Each dataset represents an area of an ellipse with two standard deviations in the anteroposterior and lateral planes about a mean point, taken over a period of 30 seconds. The resulting Kanegaonkar "K" value (200000 and - 15000) gives information about postural oscillation. For the experimental procedure, the participants will be asked to stand upright with their arms by their sides. Postural sway will be initially assessed in a normal clinic room in 1 of the 8 standing test conditions (4 different standing conditions: (1) feet shoulder wide apart, (2) feet together, (3) tandem position (4) on foam with shoulder wide apart and 2 different visual conditions: (1) eyes open, (2) eyes closed).

CONTACTS AND LOCATIONS:
Overall Officials: Betül Fatma Bilgin, PT, Principal Investigator — Eastern Mediterranean University; Gözde İyigün, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Eyalet/Yerleşke, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schoene D, Delbaere K, Lord SR. Impaired Response Selection During Stepping Predicts Falls in Older People-A Cohort Study. J Am Med Dir Assoc. 2017 Aug 1;18(8):719-725. doi: 10.1016/j.jamda.2017.03.010. Epub 2017 May 16. PMID 28526585
- [Background] Faria CA, Alves HVD, Charchat-Fichman H. The most frequently used tests for assessing executive functions in aging. Dement Neuropsychol. 2015 Apr-Jun;9(2):149-155. doi: 10.1590/1980-57642015DN92000009. PMID 29213956
- [Background] Iyigun G, Kirmizigil B, Angin E, Oksuz S, Can F, Eker L, Rose DJ. The reliability and validity of the Turkish version of Fullerton Advanced Balance (FAB-T) scale. Arch Gerontol Geriatr. 2018 Sep-Oct;78:38-44. doi: 10.1016/j.archger.2018.05.022. Epub 2018 Jun 4. PMID 29886283
- [Derived] Bilgin BF, Iyigun G. Multitask Versus Multicomponent Training on Cognitive and Motor Functions in Persons With Mild Cognitive Impairment: A Randomized Trial. J Aging Phys Act. 2022 Apr 20;30(6):1024-1037. doi: 10.1123/japa.2021-0408. Print 2022 Dec 1. PMID 35453122